CLINICAL TRIAL: NCT07289243
Title: RANDOMIZED CLINICAL TRIAL COMPARING TRANSURETHRAL PROSTATE RESECTION (TURP) AND ECHOLASER SORACTELITE-TPLA (TRANSPERINEAL LASER ABLATION) IN PATIENTS WITH LOWER URINARY TRACT SYMPTOMS DUE TO BENIGN PROSTATIC OBSTRUCTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Principal Investigator, Pasquale Ditonno, MD, Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TPLA-2023
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: RANDOMIZED
MeSH Terms: interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPLA (Other): Patients underwent TPLA tretment
  Interventions: Procedure: ECHOLASER-TPLA
- TURP (Other): Patients underwent TURP tretment
  Interventions: Procedure: TURP

INTERVENTIONS:
Procedure: ECHOLASER-TPLA — transperineal laser ablation of prostatic adenoma, by transrectal ultrasound guide.
  Other Names: TPLA
  Arms: TPLA
Procedure: TURP — Transurethral resection of prostate, by uretrocistoscopy approach.
  Arms: TURP

SUMMARY:
THIS STUDY IS A RANDOMIZED CLINICAL TRIAL COMPARING TRANSURETHRAL PROSTATE RESECTION (TURP) AND ECHOLASER SORACTELITE-TPLA (TRANSPERINEAL LASER ABLATION) IN PATIENTS WITH LOWER URINARY TRACT SYMPTOMS DUE TO BENIGN PROSTATIC OBSTRUCTION. THE PRIMARY GOAL IS TO SHOW THE NON-INFERIORITY OF TPLA VERSUS TURP BY IPSS-SCORE.

ELIGIBILITY:
Inclusion Criteria:

* age, Lower urinary tract simptoms (IPSS >= 8), uncompliance or no achived drugs treatment for IPB, prostate volume 40ml-80ml , ability to express informed consent.

Exclusion Criteria:

* previous surgical tretment for IPB, bladder catheter, bladder stones, urinary or seminal infections, hypo-/a-contractilitis of bladder, bladder tuomrs, urethral stricture, neurological bladder, refuse to sign informed consent

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 80 (Estimated)
Dates: Start 2024-07-14 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
IS TO SHOW THE NON-INFERIORITY OF TPLA VERSUS TURP BY IPSS-SCORE | one, three, six, twelve mounth after treatment

SECONDARY OUTCOMES:
COMPARE Q-MAX UROFLOW | one, three, six, twelve mounth after treatment
COMPARE INPATIENT-TIMING | one, three, six, twelve mounth after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Urologia e Trapianti di Rene Policlinico di Bari, Bari, ITALY/Bari, Italy